CLINICAL TRIAL: NCT00000461
Title: Harvard Atherosclerosis Reversibility Project (HARP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 50; R01HL036392 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Pravastatin; Niacin; Cholestyramine Resin; Gemfibrozil; Fatty Acids, Omega-3

INTERVENTIONS:
Drug: pravastatin
Drug: niacin
Drug: cholestyramine
Drug: gemfibrozil
Drug: fatty acids, omega-3

SUMMARY:
To determine by sequential coronary arteriography whether a lipid-lowering diet with and without lipid-lowering drugs could reverse coronary artery disease in normocholesterolemic patients. Also, to test whether fish oil supplements could improve human coronary atherosclerosis. Finally, to determine the effect of combination therapy with lipid-reducing drugs in patients with coronary heart disease and "normal" cholesterol levels. At least three clinical trials were conducted.

DETAILED DESCRIPTION:
BACKGROUND:

The prognosis of patients with coronary heart disease is closely related to the degree of coronary luminal obstruction. In population studies, the incidence and severity of coronary atherosclerosis on angiography is correlated with diet and plasma lipoprotein cholesterol. Previous clinical trials had shown that treatments that lowered plasma concentrations of low density lipoprotein cholesterol benefited some hypercholesterolemic patients with coronary heart disease. No similar benefit had been demonstrated in normocholesterolemic patients who make up the majority of patients with coronary heart disease.

DESIGN NARRATIVE:

In the cholesterol-lowering agent trial, all patients received Step 1 dietary instruction before randomization and every three months thereafter. Randomization was stratified by medical or surgical treatment for coronary disease and the ratio of total to HDL cholesterol. A total of 39 patients were assigned to placebo and 40 to active treatment with pravastatin, nicotinic acid, cholestyramine, and gemfibrozil stepwise as needed to reach the specified goal (total cholesterol less than or equal to 4.1 mmol/L, ratio of LDL/HDL cholesterol less than or equal to 2.0). Lipid concentrations were measured every six weeks. Baseline angiograms were compared to angiograms taken at 30 months.

In the fish oil trial, 41 patients were randomized to fish oil capsules containing 6 grams of n-3 fatty acids daily and 39 patients were randomized to olive oil placebo capsules for an average duration of 28 months. Each fish oil capsule contained 500 mg of n-3 polyunsaturated fatty acids composed of 240 mg of eicosapentaenoic acid, 160 mg of docosahexaenoic acid, and 100 mg of mainly docosapentaenoic acid. Randomization was stratified by medical or surgical treatment for coronary disease and the ratio of total to HDL cholesterol. The primary outcome variable was change in minimal diameter of coronary artery lesions expressed as a continuous variable. During the initial hospital stay for catheterization, dietary instruction was provided to every patient according to the National Cholesterol Education Program (NCEP) Step 1 guidelines. A seven-day diet record was collected at the randomization visit and every three months during the trial. Every twelve weeks, a research nurse reviewed with the patients side effects, diet, and concomitant medications and performed a pill count. Every 24 weeks, the patients received an interval medical history and physical examination by a physician. A fasting blood sample was obtained for lipid analysis at the 12- and 24-week visits and every 24 weeks thereafter. If the total cholesterol level of any patient increased to 250 mg/dl (6.43 mmol/liter) or greater on two consecutive measurements, intensified dietary instruction was given, followed by drug therapy with cholestyramine or nicotinic acid or both as needed to lower total cholesterol to less than 250 mg/dl. Twenty-one patients did not complete the protocol due to death, refusal to undergo the second cardiac catheterization, development of medical conditions precluding participation, intolerance to the capsules, and a missing initial angiogram.

In the combination therapy trial, patients were randomized to usual care or to stepped-care drug therapy with lipid-lowering agents including pravastatin, nicotinic acid, cholestyramine, and gemfibrozil to decrease total cholesterol levels to less than 160 mg/dl and the ratio of low density lipoprotein cholesterol to high density lipoprotein cholesterol to less than 2.0. Measurements included fasting serum lipoprotein profile, fasting apolipoprotein levels, and frequency of adverse effects. Patients were assessed every six weeks during drug titration and every three months thereafter for two -and-a-half years.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Men and women, normocholesterolemic, with 30 percent or greater narrowing of a coronary artery lumen as revealed by angiography. (Cholesterol-Lowering Agent Trial).

Men and women with angiographically-documented coronary heart disease (Fish Oil Tr

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1986-12; Study Completion 1992-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Sacks — Brigham and Women's Hospital

REFERENCES:
- [Background] Sacks FM, Pasternak RC, Gibson CM, Rosner B, Stone PH. Effect on coronary atherosclerosis of decrease in plasma cholesterol concentrations in normocholesterolaemic patients. Harvard Atherosclerosis Reversibility Project (HARP) Group. Lancet. 1994 Oct 29;344(8931):1182-6. doi: 10.1016/s0140-6736(94)90506-1. PMID 7934538
- [Background] Sacks FM, Stone PH, Gibson CM, Silverman DI, Rosner B, Pasternak RC. Controlled trial of fish oil for regression of human coronary atherosclerosis. HARP Research Group. J Am Coll Cardiol. 1995 Jun;25(7):1492-8. doi: 10.1016/0735-1097(95)00095-l. PMID 7759696
- [Background] Sacks FM, Gibson CM, Rosner B, Pasternak RC, Stone PH. The influence of pretreatment low density lipoprotein cholesterol concentrations on the effect of hypocholesterolemic therapy on coronary atherosclerosis in angiographic trials. Harvard Atherosclerosis Reversibility Project Research Group. Am J Cardiol. 1995 Sep 28;76(9):78C-85C. doi: 10.1016/s0002-9149(99)80475-5. PMID 7572692
- [Background] Pasternak RC, Brown LE, Stone PH, Silverman DI, Gibson CM, Sacks FM. Effect of combination therapy with lipid-reducing drugs in patients with coronary heart disease and "normal" cholesterol levels. A randomized, placebo-controlled trial. Harvard Atherosclerosis Reversibility Project (HARP) Study Group. Ann Intern Med. 1996 Oct 1;125(7):529-40. doi: 10.7326/0003-4819-125-7-199610010-00001. PMID 8815751